CLINICAL TRIAL: NCT05493371
Title: Feasibility Study of Empagliflozin As Treatment for Idiopathic Pulmonary Arterial Hypertension
Brief Title: Empagliflozin in Pulmonary Arterial Hypertension
Acronym: Emphower PoC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Harm Jan Bogaard, Prof. Dr., VU University of Amsterdam
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 81866; 2022-002400-20 (EudraCT Number); 2022-501512-33-00 (Other: Clinical Trials Information System (CTIS) EU CT Number)
Record Dates: First submitted 2022-07-28; First posted 2022-08-09 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Idiopathic Pulmonary Arterial Hypertension
Keywords: Empagliflozin
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: prospective single-center, phase IIa, single arm, open label, interventional proof-of-concept study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Empagliflozin (Experimental)
  Interventions: Drug: Empagliflozin 10 MG

INTERVENTIONS:
Drug: Empagliflozin 10 MG — 10 mg once daily empagliflozin oral tablets for 12 weeks

SUMMARY:
The aim of the study is to determine whether conducting a randomized placebo-controlled clinical trial is feasible, safe for the patient and whether the treatment is well tolerated in patients with idiopathic pulmonary arterial hypertension.

DETAILED DESCRIPTION:
This study is designed as a prospective, single-center, phase IIa, single-arm, open-label, interventional proof-of-concept trial in patients diagnosed with idiopathic pulmonary arterial hypertension (IPAH) who are currently on stable therapy. Patients will be administered a once-daily oral dose of 10 mg empagliflozin for a duration of 12 weeks along with standard treatment. The primary objective of this study is to assess safety and tolerability of empagliflozin and to assess whether a potential future randomized, double-blind, placebo-controlled study is feasible.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Diagnosis of idiopathic PAH
3. Documented diagnostic right heart catheterization (RHC) at any time prior to screening confirming diagnosis of WHO diagnostic pulmonary hypertension Group I: PAH with subtype idiopathic PAH. The documented RHC shows all of the following criteria:

   1. mPAP > 20 mmHg at rest
   2. Pulmonary artery wedge pressure (PAWP) or left ventricular end-diastolic pressure (LVEDP) ≤ 15 mmHg at rest
   3. PVR ≥ 240 dyn·sec/cm5 (3 Wood units) at rest
4. Symptomatic pulmonary hypertension classified as World Health Organization (WHO) functional class (FC) II, III or IV
5. PAH therapy is at stable (per investigator) dose levels of standard of care (SoC) therapies for at least 90 days prior screening. SoC therapy refers to a therapy consisting of at least 1 agent from a list including: an endothelin-receptor antagonist (ERA), a phosphodiesterase 5 (PDE5) inhibitor, a soluble guanylate cyclase stimulator, and/or a prostacyclin analogue or receptor agonist (SC/inhaled/PO).

Exclusion Criteria:

1. Any subject who received any investigational medication within 1 month prior to the start of this study or who is scheduled to receive another investigational drug during the course of this study. Patients participating in a purely observational trial will not be excluded
2. Females of childbearing potential, defined as a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy or 2) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 months), unable or unwillingly to either:

   1. Use highly effective methods of birth control according to the International Conference on harmonisation of pharmaceuticals for human use (ICH) that result in a low failure rate of less than 1% per year when used consistently and correctly 43. Highly effective methods include hormonal contraception (for example, birth control pills, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation (having your tubes tied); or a partner with a vasectomy who has completed follow-up to confirm a successful procedure
   2. Have a negative pregnancy tests as verified by the investigator prior to starting study therapy and agrees to have an extra pregnancy test 8 weeks after start of the study
3. Contraindication for CMR imaging as defined in the protocol of the Amsterdam UMC "Kwaliteitsdocument Cardiale MRI (Versie 1)". The list of contra-indications includes: claustrophobia, ferromagnetic implants, implanted cardioverter defibrillator (ICD) or pacemaker (except for the MR conditional) and ball-in-cage mechanic heart valve.
4. Impaired renal function, defined as eGFR < 30 mL/min/1.73 m2 (CKD-EPI) or requiring dialysis
5. History of chronic severe (Child Pugh classification score >10, Appendix 1) or active liver disease defined as serums transaminases >5 x upper limit of normal (ULN) or bilirubin > 1.5 x ULN
6. History of ketoacidosis
7. Known allergy, intolerance or hypersensitivity to empagliflozin or other SGLT-2 inhibitors
8. Use of lithium compounds and being unable or unwillingly to increase the monitoring frequency of lithium levels
9. Current or scheduled use of the following Uridine glucuronosyltransferase (UGT) inducers: phenytoin, rifampicin, carbamazepine, lamotrigine, ritonavir, efavirenz, tipranavir, phenobarbital, testosterone propionate and nelfinavir.
10. Current or prior use of a SGLT-2 inhibitor
11. Heart transplant recipient or listed for heart transplant
12. Chronic pulmonary disease requiring home oxygen or steroid maintenance therapy
13. Symptomatic hypotension and/or a systolic blood pressure (SBP) < 90 mmHg at screening
14. Gastrointestinal (GI) surgery or GI disorder that could interfere with absorption of trial medication in the investigator's opinion
15. Presence of any other disease than pulmonary arterial hypertension with a life expectancy of <1 year in the investigator's opinion
16. Women who are pregnant, nursing, or who plan to become pregnant while in the trial
17. History of severe (previously required or prolonged patient hospitalization, resulted in persistent or marked disability/incapacity) or recurrent (≥2 infections in six months or ≥3 infections in one year) genital infections.
18. History of severe hypoglycaemia (<40 - 30 mg/dL = <2.2 - 1.7 mmol/L), previous hospitalisation for hypoglycaemia or seizures attributed to hypoglycaemia
19. Active solid or haematological malignancy, with the exception of fully excised or treated basal cell carcinoma, cervical carcinoma in-situ, or ≤ 2 squamous cell carcinomas of the skin
20. History or suspicion of inability to cooperate adequately
21. Any condition that, in the investigator's opinion, makes them an unreliable trial subject or unlikely to complete the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Tolerability: the number of patients who have to prematurely discontinue treatment due to intolerability or adverse events. | 12 weeks
Feasibility: time needed to include all patients and number of patients needed to screen. | 12 weeks
Safety: the number of adverse events (AEs), severe adverse events (SAEs), adverse event of special interest (AESI) and suspected unexpected serious adverse reactions (SUSARs). | 12 weeks

SECONDARY OUTCOMES:
Right ventricle ejection fraction (RVEF) measured using MRI | 12 weeks
  RVEF is calculated using the RVESV, RVEDV
Right ventricle mass measured using MRI | 12 weeks
Left ventricle ejection fraction (LVEF) measured using MRI | 12 weeks
  LVEF is calculated using the LVESV, LVEDV
Stroke volume (SV) measured using MRI | 12 weeks
  SV is calculated using the LVESV, LVEDV
Tricuspid annular plane systolic excursion (TAPSE) measured using transthoracic ultrasound | 12 weeks
Estimated sPAP measured using transthoracic ultrasound | 12 weeks
Right ventricle fractional area change (RVFAC) measured using transthoracic ultrasound | 12 weeks
Blood biomarkers | 12 weeks
  Endpoints: Expression of peroxisome proliferator-activated receptor gamma coactivator 1-alpha (PGC-1α) and bone morphogenetic protein receptor II (BMPR2) in peripheral blood mononuclear cells (PMBC)
Blood safety biomarkers | 12 weeks
  Fasting glucose, N-terminal prohormone of Brain Natriuretic Peptide (NT-proBNP) and creatinine in blood.
Urine safety biomarkers | 12 weeks
  Ketones, nitrites, leukocytes and glucose in urine test strip (dipstick).
Functional class | 12 weeks
  World Health Organization Function Classification of Pulmonary Hypertension. Outcome: Class I, Class II, Class III or Class IV
Six-Minute Walk Distance | 12 weeks
  Six-minute walk distance (6MWD) will be measured by the 6-minute walk test (6MWT). The test should preferably be conducted on a straight 30 metre track. The patient is instructed to walk as far as possible for six minutes. One lap is demonstrated. The patient is told that slowing down can be necessary, and after pausing are encouraged to start walking as soon as possible.
Quality of life measured with use of the EMPHASIS-10 questionnaire | 12 weeks
  The emPHasis-10 is a short questionnaire for assessing Health-related quality of life in pulmonary arterial hypertension. The questionnaire comprises 10 items that are formatted as a semantic six-point differential scale and results in a score out of 50 where a higher score represents a higher symptom burden.
Quality of life measured with use of the Cambridge Pulmonary Hypertension Outcome Review (CAMPHOR) questionnaire | 12 weeks
  The CAMPHOR questionnaire contains 65 items in total. The measure consists of three different scales: a symptom scale assessing energy, breathlessness and mood (25-items; low score indicating minimal symptoms); activity limitations scale with a 3-point rating system (15-items; range 0 to 30, lower score indicating minimal activity limitation); and a QoL scale (25-items; lower score indicating better QoL). It is negatively weighted; a higher score indicates worse QoL and greater functional limitation.

CONTACTS AND LOCATIONS:
Overall Officials: Harm Jan Bogaard, Prof. dr., Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- Amsterdam UMC, location Vumc, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
On reasonable request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Six months after study completion
Access Criteria: data can be obtained on request by email